CLINICAL TRIAL: NCT06932185
Title: Transcranial Ultrasound to Disrupt Pathological Oscillations in the Brain of People With Parkinson's Disease and Other Neurological Disorders
Brief Title: TUS to Disrupt Pathological Oscillations
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 322261
Record Dates: First submitted 2025-03-27; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TUS active (Experimental)
  Interventions: Other: Transcranial Focussed Ultrasound - Active
- TUS sham (Sham Comparator)
  Interventions: Other: Transcranial Focussed Ultrasound - Sham
- TUS Active Control (Active Comparator)
  Interventions: Other: Transcranial Focussed Ultrasound - Active control

INTERVENTIONS:
Other: Transcranial Focussed Ultrasound - Active — Transcranial focussed ultrasound to target site
  Arms: TUS active
Other: Transcranial Focussed Ultrasound - Sham — Transcranial focussed ultrasound off
  Arms: TUS sham
Other: Transcranial Focussed Ultrasound - Active control — Transcranial focussed ultrasound on to control
  Arms: TUS Active Control

SUMMARY:
Scientists and clinicians are interested in measuring and perturbing the signals in the brain - both to better understand normal operation and explore new therapy options for disease. One example of a signal is a "brainwave," also called a neural oscillation, which is a periodic oscillation of the electrical signals in the brain and which are linked to both normal and abnormal brain function.

When circuits in the brain are not working properly, investigators can see changes in the characteristics of these oscillations. Many neurological conditions produce changes in brainwaves. For example, in patients with Parkinson's disease, oscillations in the "beta band" (approximately 15Hz) are observed to be more prominent. In another example, investigators see similar large oscillations in the presence of a seizure in people with epilepsy. Disrupting these abnormal oscillations can treat some of the symptoms of disease. One example of this is found in Parkinson's disease, where surgeons can implant electrodes deep in the brain and electrically stimulate cells by a process called deep brain stimulation (DBS). With DBS, it is possible to suppress these beta oscillations and improve symptoms. However, DBS is a highly invasive procedure that includes the need for a burr hole in the skull, placement of the electrode in the brain, and insertion of a "pacemaker" in the chest with wires tunnelled through the neck. The investigators propose to use ultrasound to modify pathological brainwaves non-invasively.

While the proof-of-concept is in Parkinson's disease, the potential impact is much broader - if successful, the investigators will provide a non-invasive paradigm for probing the brain and exploring novel treatments for neurological conditions, such as pain and cognitive disorders.

DETAILED DESCRIPTION:
Transcranial Ultrasound Stimulation (TUS):

TUS will be applied using a commercially available transcranial ultrasound transducer and neuronavigation system that allows for targeting of specific brain regions. TUS targeting will be based on participant specific MRI and CT scans that take place as part of routine pre-operative planning before DBS implantation. TUS will then be applied during cognitive and motor tasks as described below.

Clinical assessments:

During each step of the study visit, during TUS to each target, clinical assessments will be made for each participant. These will be specific to the disease of interest and will be completed by a clinician. They will be filmed so that they can be assessed by blinded assessors after the study visit and allow for blinded quantification of TUS on clinical symptoms. A member of the research team will film assessments whilst a clinician completes them, and they will later scramble the video files to allow blinded assessment at a later date.

Cognitive tasks include a dot direction discrimination task and for pain participants will include quantitative sensory testing. Motor tasks will include a stop signal task.

During the TUS, Sham and Alternative brain target TUS, measurements will include EEG, Local Field Potentials (LFPs) recorded from the DBS electrodes, ECG.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Implanted Medtronic Percept or equivalent DBS system (one that can measure LFPs) or externalised depth electrodes as part of routine care
* Participant willing and able to tolerate transcranial ultrasound stimulation.
* Stable therapy with no drug changes in past 6 weeks
* Measurable beta peak on screening

Exclusion Criteria:

* Patients with extreme language barrier that cannot understand the purpose or instructions of the study despite the use of an interpreter.
* Patients with implanted electrodes without telemetric capacity.
* Co-morbid neurological disorder that may confound results, e.g. second motor impairment.
* Fever at time of study visit (>38 degrees Celsius)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2028-06-09 (Estimated); Study Completion 2028-07-09 (Estimated)

PRIMARY OUTCOMES:
LFP modulation | Change from baseline during ultrasound
  Electrical activity recorded from indwelling Deep Brain Stimulation electrodes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided